CLINICAL TRIAL: NCT04838418
Title: Transorbital Ultrasound and Other Markers for Prognosis Prediction After Cardiac Arrest (TOMCAT)
Brief Title: Transorbital Ultrasound and Other Markers for Prognosis Prediction After Cardiac Arrest
Acronym: TOMCAT
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital Pilsen (Other)
Collaborators: Na Homolce Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TOMCAT
Record Dates: First submitted 2021-04-06; First posted 2021-04-09 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — microRNA, copeptine and NSE sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Optic nerve sheath diameter measured by transorbital ultrasound — Optic nerve sheath diameter measured 3 mm behind eyeball. For every eyeball 2 measurements in axial and 2 measurements in sagital projections are performed. Summary value for every eyeball is arithmetic mean from these 4 measurements.

SUMMARY:
In sudden cardiac arrest patients with return of spontaneous circulation, brain damage is one of the main determinants of short-term mortality and poor prognosis (CPC 3-5). It is important to properly select group of patients in whom treatment is futile. According to current guidelines, multimodal approach is recommended. Optic nerve sheath diameter measured by ultrasound is non-invasive, fast, low-cost and readily available bed-side method, but evidence for its use as neuroprognostication modality is limited to only few small studies. The aim of this study is to evaluate validity of ONSD as neuroprognostication method at larger cohort of patients, compare it with other established methods and compare ultrasound and CT measurement of ONSD.

DETAILED DESCRIPTION:
Additional relevant MeSH terms:

cardiac arrest, cardiovascular diseases, optic nerve sheath diameter.

ELIGIBILITY:
Inclusion Criteria:

* age of 18 years or older
* out of hospital cardiac arrest of non-traumatic cause with CPR and subsequent ROSC
* Glasgow coma scale (GCS) ≤ 7 or sedation 30 minutes after ROSC achievment

Exclusion Criteria:

* unavailable first measurment of the optic nerve sheath diameter (ONSD) measured by transorbital ultrasonography 24±6 hours after ROSC achievement
* refractory cardiac arrest
* craniocerebral injury
* intracranial tumor
* active intracranial bleeding
* haemorrhagic stroke and/or subarachnoid haemorrhage in the last 3 months
* facial trauma affecting the eye area
* active neuroendocrine tumor, small cell lung cancer, non-small cell lung
* CPC 3-5 before cardiac arrest
* sclerosis multiplex and/or optic neuritis of other etiology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients after cardiac arrest with subsequent ROSC, 18 years of age and older
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Value of ONSD for short-term neurological outcome prediction | 30 days
  Assessment of the correlation between the optic nerve sheath diameter measured by transorbital ultrasonography and neurological outcome of patients (quantified by the CPC scale) after out of hospital cardiac arrest with subsequent ROSC
Value of ONSD for short-term mortality prediction | 30 days
  Assessment of the correlation between optic nerve sheath diameter measured by transorbital ultrasonography and mortality during a 30-day follow-up.

SECONDARY OUTCOMES:
Comparison of ONSD and electrophysiologic modalities for neurological outcome prediction | 96 hours
  Assessment of the correlation between the optic nerve sheath diameter measured by transorbital ultrasonography and negative prognostic markers obtained by somatosensory evoked potentials examination and EEG in patients remaining in a coma even after the end of therapeutic hypothermia and sedation.
Comparison of ONSD measurements by ultrasonography and computed tomography | 48 hours
  Assessment of accuracy of the optic nerve sheath diameter measured by ultrasonography compared to CT measurement performed 48 ± 12 hours after achievment of ROSC.
Correlation between ONSD and fundoscopic signs of papillary edema | 48 hours
  Assessment of the correlation between the optic nerve sheath diameter measured by transorbital ultrasonography and grade of optic nerve papillary edema quantified by the Frisen scale on fundoscopic examination performed 48 ± 12 hours after achievment of ROSC.
Correlation between ONSD and thickness of retinal nerve fibers measured by OCT | 5 months
  Assessment of the correlation between the optic nerve sheath diameter measured by transorbital ultrasonography and thickness of retinal nerve fibers measured by optical coherence tomography at time intervals of 1, 3 and 5 months after achievment of ROSC.
Effect of blood carbon dioxide on ONSD | 72 hours
  Assessment of the correlation between the optic nerve sheath diameter measured by transorbital ultrasonography and paCO2 and ETCO2 values at the time of measurement.
Value of ONSD for long-term neurological outcome and mortality | 6 months
  Assessment of the correlation between the optic nerve sheath diameter measured by transorbital ultrasonography and mortality and neurological outcome of patients (quantified by the CPC scale) at 6 months after ROSC.
Correlation between blood NSE, copeptin and selected RNAs | 6 months
  Assessment of the correlation between blood NSE, copeptin and selected micro-RNAs measured at defined time intervals from ROSC, to neurological outcome prediction in patients after out of hospital cardiac arrest with subsequent ROSC.

CONTACTS AND LOCATIONS:
Overall Officials: Štefan Volovár, MUDr., Principal Investigator — University hospital Plzen
Locations (1):
- University Hospital Plzen, Pilsen, Czechia

IPD SHARING:
Plan to Share IPD: No